CLINICAL TRIAL: NCT01489527
Title: Preparedness Study: Efficacy of HPV Vaccine to Reduce HIV Infection
Brief Title: Preparedness Study - HPV Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MCC-16685; IISP ID 39582 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-01

CONDITIONS: Sexual Transmission of Infection
Keywords: Vaccine; Placebo; sexually transmitted infection (STI); HIV; Human Immunodeficiency; Gardasil; HPV; human papillomavirus
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gardasil Vaccine Administration (Active Comparator): Gardasil Vaccine Administration. Family Health International (FHI) statisticians randomly assigned each participant an allocation number and then subsequently assigned a unique vial identification number for the vial of vaccine the participant should receive at each visit. A single participant could not be assigned more than 1 allocation number.
  Interventions: Biological: Gardasil Vaccine
- Placebo Administration (Placebo Comparator): Placebo Administration. Family Health International (FHI) statisticians randomly assigned each participant an allocation number and then subsequently assigned a unique vial identification number for the vial of vaccine the participant should receive at each visit. A single participant could not be assigned more than 1 allocation number.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Gardasil Vaccine — The study vaccine was blindly administered as supplied on Day 1, Month 2, and Month 6. All vaccines were injected intramuscularly into the deltoid muscle by a member of the clinical staff.
  Other Names: Gardasil
  Arms: Gardasil Vaccine Administration
Other: Placebo — The study vaccine was blindly administered as supplied on Day 1, Month 2, and Month 6. All vaccines were injected intramuscularly into the deltoid muscle by a member of the clinical staff.
  Arms: Placebo Administration

SUMMARY:
Moffitt Cancer Center is the Coordinating Center for this study.

The purpose of this study is to develop and test the infrastructure to conduct a future Phase III vaccine efficacy trial to assess trial feasibility, and to assess human papillomavirus (HPV) genotype distribution, data needed to design a Phase III trial. The investigators propose to conduct a Preparedness study among women ages 16-24 years of age residing in a region of South Africa with a high human immunodeficiency (HIV) incidence and prevalence.

The specific aims of this study are to:

1. Identify, recruit, enroll, and randomize a cohort of HIV negative women (200 per arm, 400 total) ages 16-24 years to an HPV vaccine against 4 types (HPV 6, 11, 16, 18 [Gardasil]) or placebo vaccine.
2. Determine the cervical HPV prevalence and type distribution at enrollment, and cervical lesion prevalence among young females ages 16-24 years at high risk for HIV infection.
3. Assess the rate of compliance through the 3-dose vaccination series

DETAILED DESCRIPTION:
The study vaccine will be blindly administered as supplied on Day 1, Month 2, and Month 6. Both HPV and placebo vaccines will be in identical bottles, and all treatment codes will be kept under lock and key. All vaccines will be injected intramuscularly into the deltoid muscle by a member of the clinical staff. Each participant will be monitored for systemic and local reactions for 30 minutes postvaccination after each study vaccination for any adverse effects, including allergic reactions. Vaccine adverse events will continue to be monitored throughout the duration of the study period. Vaccine will be shipped to a central pharmacy at Stellenbosch University and stored in a refrigerator monitored and maintained at 2-8 C prior to distribution and local storage at participating clinical centers.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 16-24 years of age residing in a region of South Africa with a high HIV incidence and prevalence
* HIV negative
* has ever had vaginal intercourse
* has never had Papanicolaou smear (Pap) testing or has only had normal Pap test results
* fully understands study procedures, risks involved in the study, and voluntarily agrees to participate by giving written informed consent
* agrees to refrain from douching/vaginal cleansing and using vaginal medications or preparations for 2 calendar days prior to the Day 1 visit as well as other future visits that include collection of cervical specimens
* agrees to refrain from sexual intercourse for 2 calendar days prior to the Day 1 visit as well as other future visits that include collection of cervical specimens
* agrees to utilize effective contraception during sexual intercourse (excluding the rhythm method, withdrawal alone, and emergency contraception) during the vaccination period.
* Informed consent procedures for females <18 years of age: Informed consent and informed assent will be obtained from parents/legal guardians and adolescents respectively, prior to participation. The consent form will include information about the study and individual request for consent of participants to participate in the study. It will be emphasized that participation is voluntary and that participants are free to withdraw from the study at any stage without any disadvantage to them. An assessment of understanding will be conducted at screening to ensure that consent is informed.

Exclusion Criteria:

* have a history of severe allergic reaction
* have a known allergy to any vaccine component (e.g., aluminum, yeast, or BENZONASE)
* are currently immuno-compromised
* have received a marketed HPV vaccine, or are pregnant and lactating

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 406 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Giuliano, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States
- Stellenbosch University, Parow, South Africa, South Africa

REFERENCES:
- [Derived] Menezes LJ, Pokharel U, Sudenga SL, Botha MH, Zeier M, Abrahamsen ME, Glashoff RH, Engelbrecht S, Schim van der Loeff MF, van der Laan LE, Kipping S, Taylor D, Giuliano AR. Patterns of prevalent HPV and STI co-infections and associated factors among HIV-negative young Western Cape, South African women: the EVRI trial. Sex Transm Infect. 2018 Feb;94(1):55-61. doi: 10.1136/sextrans-2016-053046. Epub 2017 May 10. PMID 28490581
- [Derived] Sudenga SL, Torres BN, Botha MH, Zeier M, Abrahamsen ME, Glashoff RH, Engelbrecht S, Schim Van der Loeff MF, Van der Laan LE, Kipping S, Taylor D, Giuliano AR. HPV SEROSTATUS PRE- AND POST-VACCINATION IN A RANDOMIZED PHASE II PREPAREDNESS TRIAL AMONG YOUNG WESTERN CAPE, SOUTH AFRICAN WOMEN: THE EVRI TRIAL. Papillomavirus Res. 2017 Jun;3:50-56. doi: 10.1016/j.pvr.2017.02.001. Epub 2017 Feb 16. PMID 28480334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women residing in the Western Cape, South Africa were enrolled from November 2012 to July 2013 in a preparedness study. Participants were recruited from the Kraaifontein day hospital and the Bloekombos primary health care clinic by community workers and through word of mouth, flyers, and brochures.
Pre-assignment Details: 4 of the 406 participants randomized had a false HIV negative test result, reducing the participants to 202 in the Gardasil Arm and 200 in the Placebo Arm.
Groups:
- Gardasil Vaccine Administration: Gardasil Vaccine injected intramuscularly into the deltoid or thigh muscle.
- Placebo Administration: Placebo injected intramuscularly into the deltoid or thigh muscle.
Period: Overall Study
Arm/Group | Gardasil Vaccine Administration | Placebo Administration
Started | 205 | 201
Completed | 183 | 175
Not Completed | 22 | 26
Not completed — Pregnancy | 9 | 14
Not completed — Participant moved | 6 | 7
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Lost to Follow-up | 5 | 1
Not completed — Procedures | 1 | 0
Not completed — Not compliant | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Gardasil Vaccine Administration | Placebo Administration | Total
Number analyzed (Participants) | 202 | 200 | 402
Age, Continuous [Median (Full Range); unit: years] | 20 [16 to 24] | 20 [16 to 24] | 20 [16 to 24]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 46 | 86
  Between 18 and 65 years | 162 | 154 | 316
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 200 | 402
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 202 | 200 | 402

OUTCOME MEASURES:

1. Primary Outcome: Human Papillomavirus (HPV) Rate
Description: HPV type distribution and prevalence of each HPV type at enrollment.
Time Frame: At Enrollment - 5 Month Enrollment Period
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Gardasil Vaccine Administration | Placebo Administration
Number analyzed (Participants) | 202 | 200
participants
  Any HPV Type | 143 | 136
  Any High-Risk Type | 106 | 113
  Any Low-Risk Type | 103 | 97
  HPV6 | 9 | 3
  HPV11 | 2 | 2
  HPV16 | 23 | 32
  HPV18 | 11 | 14

2. Secondary Outcome: Study Compliance Rate
Description: Percentage of participants to complete the 3-dose vaccination series and all 4 study visits.
Time Frame: 18 Months
Population: All treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Gardasil Vaccine Administration | Placebo Administration
Number analyzed (Participants) | 202 | 200
percentage of participants | 91.5 | 87.5

3. Secondary Outcome: Percentage of Participants Who Were Seropositive by HPV Type
Description: Percentage of participants who were seropositive to HPV at enrollment, by specific HPV type.
Time Frame: At Enrollment - 5 Month Enrollment Period
Population: All treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Gardasil Vaccine Administration | Placebo Administration
Number analyzed (Participants) | 202 | 200
percentage of participants
  HPV6 | 73 | 73
  HPV11 | 45 | 47
  HPV16 | 32 | 37
  HPV18 | 46 | 41
  HPV31 | 31 | 38
  HPV33 | 25 | 30
  HPV45 | 15 | 18
  HPV52 | 36 | 35
  HPV58 | 36 | 36

4. Secondary Outcome: Percentage of Participants Seroconverted to HPV Types 6, 11, 16, or 18
Description: Percentage of participants who seroconverted to HPV types 6, 11, 16, or 18, following receipt of 3 doses of qHPV vaccine.
Time Frame: 18 Months
Population: Participants who were randomized to Gardasil and received all 3 doses of Gardasil
Measure: Number; unit: percentage of participants
Arm/Group | Gardasil Vaccine Administration | Placebo Administration
Number analyzed (Participants) | 179 | 0
percentage of participants | 100 |

5. Secondary Outcome: Percentage of Participants Who Seroconverted to HPV Types 31, 33, 45, or 58
Description: The percent of women that seroconverted among those receiving qHPV vaccine compared to placebo vaccine recipients for HPV types 31, 33, 45, and 58, HPV types not directly targeted by the qHPV vaccine.
Time Frame: 18 Months
Population: All treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Gardasil Vaccine Administration | Placebo Administration
Number analyzed (Participants) | 202 | 200
percentage of participants
  HPV31 | 82 | 39
  HPV33 | 56 | 34
  HPV45 | 42 | 19
  HPV58 | 69 | 38

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Arm/Group | Gardasil Vaccine Administration | Placebo Administration
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/200
Other Adverse Events (participants affected / at risk) | 59/202 | 62/200
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gardasil Vaccine Administration (N=202) | Placebo Administration (N=200)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 3 (3) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 16 (18) | 5 (5)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Immune system disorders - Other (Immune system disorders) | 2 (2) | 1 (1)
Lip infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 12 (12)
Vaginal infection (Infections and infestations) | 18 (18) | 16 (17)
Vulval infection (Infections and infestations) | 2 (2) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 5 (5)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 4 (4) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Vaginal discharge (Reproductive system and breast disorders) | 3 (3) | 5 (5)
Vaginal dryness (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The EVRI Trial had a short duration with limited follow-up time; therefore, clinical efficacy in reducing HIV acquisition cannot be assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes